CLINICAL TRIAL: NCT02040558
Title: A Multicenter, Open-Label, Phase 1 First in Human Dose Escalation Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of Intravenous MNK-010 in Subjects With Advanced Solid Tumors
Brief Title: Trial to Study the Safety of Intravenous MNK-010 in Advanced Solid Tumors
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Mallinckrodt (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: COV10100386
Record Dates: First submitted 2014-01-13; First posted 2014-01-20 (Estimated); Last update posted 2017-04-05 (Actual); Status verified 2017-04

CONDITIONS: Advanced Solid Tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- MNK-010 (Experimental): Subjects will receive 1 dose of MNK-010 followed by a 7-day post dose assessment period per treatment cycle. Dose levels will be based upon the amount of active delivered per square meter of body surface area (mg/m2). Cycles will repeat every 3 weeks (21 days) based on toxicity and response, as determined by a Safety Review Committee (SRC). Subjects will continue treatment with MNK-010 until unacceptable toxicity, documented progression of disease, another criterion for discontinuation is met, or until 4 treatment cycles have been completed.
  Interventions: Drug: MNK-010

INTERVENTIONS:
Drug: MNK-010

SUMMARY:
This is a multicenter, open-label, dose escalation study of MNK-010 in subjects with advanced solid malignancies who have failed conventional therapy. The safety, tolerability, pharmacokinetic (PK) profile, and preliminary antitumor activity of ascending doses of MNK-010 will be evaluated in subjects with advanced solid tumors.

ELIGIBILITY:
Inclusion criteria:

1. Diagnosis of an advanced solid tumor malignancy.
2. Histological or cytological evidence of malignancy.
3. Advanced malignancy, metastatic or unresectable, that has recurred or progressed following standard therapy or failed standard therapy; or for which no standard therapy currently exists, or for which subject is not a candidate for, or is unwilling to undergo, standard therapy.
4. Disease that is currently not amenable to curative surgical intervention.
5. Eastern Cooperative Oncology Group (ECOG) performance status of 0-1 and a life expectancy > 12 weeks.
6. Subject (and/or parent/guardian for subject who otherwise is unable to provide independent consent, if acceptable to and approved by the site and/or site's IRB) must be willing to give written informed consent and be able to adhere to dose and visit schedules.
7. 18 years or older, of either sex, and of any race
8. Female subjects of childbearing potential must have negative pregnancy test within 7 days prior to first dose of study drug; practicing an acceptable form of birth control for greater than 2 months prior to screening and commits to use for the duration of the study and for 3 months following the last dose of study treatment.
9. Male subjects must be sterile (biologically or surgically) or commit to the use of a reliable method of birth control for the duration of the study until at least 3 months after the last dose of study treatment in such a manner that the risk of pregnancy for a partner is minimized.
10. Prior to study treatment administration, at least 21 days must have elapsed since the subject's prior investigational or non-investigational systemic therapy, or any major surgery, and at least 21 days since prior radiotherapy.
11. Subjects with a history of prior radiotherapy are eligible if they meet the following parameters: Prior to study treatment administration, must be ≥ 21 days post-therapy and have recovered from all toxicities; must have evidence of measurable disease outside the radiation fields or radiologically confirmed progression of disease; must not have had > 25% of their functional bone marrow irradiated. Must have radiologically measureable disease, a life expectancy > 12 weeks, and adequate organ function.

Exclusion Criteria:

1. Subject has received any chemotherapy, immunotherapy, vaccines, monoclonal antibodies, whether conventional or investigational, major surgery within 21 days, or radiotherapy within 21 days of treatment in this study, or at any time during the study.
2. Subject has an active, uncontrolled systemic infection considered opportunistic, life-threatening, or clinically significant at the time of treatment.
3. Subject has symptomatic or untreated central nervous system (CNS) metastases; any type of active seizure disorder; febrile neutropenia; ≥ Grade 2 peripheral neuropathy; peritoneal or pleural effusions requiring a tap more frequently than every 14 days; QT interval corrected (QTc) prolongation or a prior history of serious arrhythmias or significant abnormalities on screening ECG; previously experienced a severe reaction to a liposomal product or a taxane; received IV treatment for bacterial/fungal infection within 7 days of screening.
4. Subject has known significant cardiovascular disease or cerebrovascular accident within 3 months of enrollment, or within the timeframe as stipulated in the additional criteria outlined in the protocol.
5. Subject requires the use of the following concomitant treatments/procedures at any time, per protocol.
6. Subject requires either moderate or strong (if weak, 2 or more) inhibitors or inducers of Cytochrome P450 3A (CYP3A) mediated metabolism.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2013-07; Primary Completion 2016-05 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) | 27 months
  MTD of MNK-010
Treatment-emergent adverse events (TEAEs) | 27 months
  Incidence of treatment-emergent adverse events (TEAEs), serious adverse events (SAEs), adverse events (AEs) of at least Grade 3 severity, and discontinuations due to AEs. AEs will be evaluated and categorized in accordance with the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events
Clinical labs | 27 months
  Changes from baseline in clinical laboratory assessments, vital signs, arterial oxygen saturation (SaO2) by pulse oximetry, physical examination, and 12-lead electrocardiograms (ECGs)

SECONDARY OUTCOMES:
Plasma PK | 27 months
  Standard plasma PK parameters will be measured following single and multiple doses.
Overall response | 27 months
  Best confirmed overall response based on Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1

CONTACTS AND LOCATIONS:
Locations (1):
- Dana Farber Cancer Institute, Boston, Massachusetts, United States